CLINICAL TRIAL: NCT02749981
Title: Cefazolin Dosing in Children Undergoing Cardiac Surgery With Cardiopulmonary Bypass
Acronym: CEFA
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/631-632-633
Record Dates: First submitted 2015-10-20; First posted 2016-04-25 (Estimated); Last update posted 2023-05-18 (Actual); Status verified 2017-05

CONDITIONS: Cardiopulmonary Bypass
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cefazolin: patients receiving cefazolin as part of routine clinical care
  Interventions: Procedure: blood and tissue sampling

INTERVENTIONS:
Procedure: blood and tissue sampling

SUMMARY:
Pharmacokinetics of cefazolin in children undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing cardiac surgery with cardiopulmonary bypass
* minimum weight 1.8 kg
* intra-arterial or intravenous access other than the drug infusion line available for blood sampling (arterial line is preferred)

Exclusion Criteria:

* no catheter in place for blood sampling
* absence of parental/patient consent
* known hypersensitivity to cefazolin

Ages: 0 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2012-12; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the time during which the unbound cefazolin concentration is above the MIC of S. aureus (fT>MIC) with the current dosing regimen | 3 years

SECONDARY OUTCOMES:
Optimalisation of the cefazolin dosing regimen to aim for a target unbound cefazolin concentration above the MIC of S. aureus during surgery | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Francois, MD, Principal Investigator — Ghent University Hospital, Department of Cardiac Surgery

REFERENCES:
- [Derived] De Cock PA, Mulla H, Desmet S, De Somer F, McWhinney BC, Ungerer JP, Moerman A, Commeyne S, Vande Walle J, Francois K, Van Hasselt JG, De Paepe P. Population pharmacokinetics of cefazolin before, during and after cardiopulmonary bypass to optimize dosing regimens for children undergoing cardiac surgery. J Antimicrob Chemother. 2017 Mar 1;72(3):791-800. doi: 10.1093/jac/dkw496. PMID 27999040